CLINICAL TRIAL: NCT04316377
Title: Norwegian Coronavirus Disease 2019 Study: An Open Labeled Randomized Controlled Pragmatic Trial to Evaluate the Antiviral Effect of Chloroquine in Adult Patients With SARS-CoV-2 Infection
Brief Title: Norwegian Coronavirus Disease 2019 Study
Acronym: NO COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Olav Dalgard, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 121446
Record Dates: First submitted 2020-03-13; First posted 2020-03-20 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Corona Virus Infection
Keywords: Corona virus infection; Chloroquine; Pragmatic trial
MeSH Terms: conditions — Coronavirus Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Two-arm, open label, pragmatic randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Chloroquine therapy in addition to standard of care
  Interventions: Drug: Hydroxychloroquine Sulfate
- No Treatment (No Intervention): Standard of care

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — 400 mg hydroxychloroquine sulphate (equalling 310 mg base) twice daily for seven days
  Other Names: Plaquenil
  Arms: Treatment

SUMMARY:
In the current proposal, the investigators aim to investigate the virological and clinical effects of chloroquine treatment in patients with established COVID-19 in need of hospital admission. Patients will be randomized in a 1:1 fashion to standard of care or standard of care with the addition of therapy with chloroquine.

DETAILED DESCRIPTION:
Chloroquine is one of two therapeutics (in addition to remdesivir) that has demonstrated in vitro inhibitory effects on SARS-CoV-2 and the drug is immediately available from national pharmacies. No delay is accordingly expected in treatment initiation after study commencement. In light of the evidence supporting chloroquine as a promising therapeutic in patients with COVID-19, the expected impact of the current proposal is considerable both in the short- and long-term. If successful, treatment with chloroquine has the potential to be the first evidence based treatment for COVID-19. The drug is affordable and the risk of side effects is low, making it an attractive therapeutic in large proportions of the population on a global scale.

In the current proposal aims to investigate the virological and clinical effects of chloroquine treatment in patients with established SARS-CoV-2 in need of hospital admission. The investigators hypothesize that early treatment with chloroquine in patients with established COVID-19 is safe and will significantly improve prognosis and impact clinical outcomes. More specifically, the investigators hypothesize that early treatment with chloroquine will increase the virological clearance rate of SARS-CoV-2, and lead to more rapid resolve of clinical symptoms, decreased proportion of patients with clinical deterioration and a decreased admission rate to intensive care units and in-hospital mortality. Considering the immediate and worldwide health emergency associated with the SARS-CoV-2 outbreak and the current lack of evidence based medical interventions for this patient group, studies investigating such possible treatment modalities in COVID-19 are direly needed.

The study is a two-arm, open label, pragmatic randomized controlled trial (RCT) designed to assess the virological and clinical effect of chloroquine therapy in patients with established COVID-19. Pragmatic clinical trials are characterized by focus on informing decision-makers on optimal clinical medicine practice and an intent to streamline procedures and data collection in the trial. By utilizing resources already paid for by the hospitals (physicians and nurses in daily clinical practice), pragmatic clinical trials can include a larger number of patients at a short time duration and at a lower cost. Due to the immediate need for study commencement and the time frame of the current proposal, a pragmatic approach will enable swift initiation of randomization and treatment. Data will be extracted from the data warehouse at Akershus University Hospital for eligible patient identification (i.e. electronic surveillance) and for automatic data extraction to the study specific database. The study will not be able to procure an acceptable placebo treatment and the study will accordingly not be placebo-controlled.

All patients at Akershus University Hospital with suspicion of acute respiratory tract infections are examined with a nasopharyngeal swab, with subsequent microbiological examination, including SARS-CoV-2 specific RT-PCR. Participants will be recruited from the entirety of the inpatients at the participating hospitals. Electronic real-time surveillance of laboratory reports from the Department of Microbiology will be examined regularly, with maximum interval 24 hours, for SARS-CoV-2 positive subjects.

The study aims to include patients by a sequential adaptive approach, where analyses are planned after the inclusion of 51 patients, with subsequent analyses after 101, 151 and 202 completed patients. All patients included in each sequence will be used for the final analyses of the entire study. This approach will enable frequent assessment of all outcome measures.

Data will be collected from the hospital electronic record system, including electronic patient records, laboratory and medical imaging systems, and prescribing systems. The data warehouse at Akershus University Hospital will be utilized for automatic data extraction to the study specific database. All clinical variables will be registered in the study eCRF system, including clinical endpoints and quantitative virological results from serial oropharyngeal specimens.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised
* Adults 18 year or older
* Moderately severe disease (NEWS score ≤ 6)
* SARS-CoV-2 positive nasopharyngeal swab
* Expected time of admission > 48 hours
* Signed informed consent must be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

* Requiring ICU admission at screening
* History of psoriasis
* Known adverse reaction to hydroxychloroquine sulphate
* Pregnancy
* Prolonged QT interval (>450 ms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
Rate of decline in SARS-CoV-2 viral load | Baseline (at randomization) and at 96 hours
  Viral load assessed by real time polymerase chain reaction in oropharyngeal samples

SECONDARY OUTCOMES:
Change in National Early Warning Score score | Baseline (at randomization) and at 96 hours
  National Early Warning Score score determines the degree of illness of a patient. Scores range from 0-20, with a higher score representing further removal from normal physiology and a higher risk of morbidity and mortality.
Admission to intensive care unit | At all times after randomization during index admission (between admission and discharge, approximately 21 days)
  Transfer from regular ward to intensive care unit during index admission
In-hospital mortality | At all times after randomization during index admission (between admission and discharge, approximately 21 days)
  All-cause mortality during index admission
Duration of hospital admission | During index admission (between admission and discharge, approximately 21 days)
  Total days admitted to the hospital (difference between admission date and discharge date of index admission)
Mortality at 30 and 90 days | At follow-up 30 and 90 days
  All-cause mortality assessed at 30 and 90 days
Clinical status | 14 days after randomization
  Percentage of subjects reporting each severity rating on a 7-point ordinal scale:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen
  6. Not hospitalized, but unable to resume normal activities
  7. Not hospitalized, with resumption of normal activities
Change in C-reactive protein concentrations | Baseline (at randomization) and at 96 hours
  Change in C-reactive protein concentrations from randomization to 96 hours after randomization
Change in alanine aminotransferase concentrations | Baseline (at randomization) and at 96 hours
  Change in alanine aminotransferase concentrations from randomization to 96 hours after randomization
Change in aspartate aminotransferase concentrations | Baseline (at randomization) and at 96 hours
  Change in aspartate aminotransferase concentrations from randomization to 96 hours after randomization
Change in bilirubin concentrations | Baseline (at randomization) and at 96 hours
  Change in bilirubin concentrations from randomization to 96 hours after randomization
Change in estimated glomerular filtration rate | Baseline (at randomization) and at 96 hours
  Change in estimated glomerular filtration rate from randomization to 96 hours after randomization
Change in cardiac troponin concentrations | Baseline (at randomization) and at 96 hours
  Change in cardiac troponin concentrations from randomization to 96 hours after randomization
Change in natriuretic peptide concentrations | Baseline (at randomization) and at 96 hours
  Change in natriuretic peptide concentrations from randomization to 96 hours after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Olav Dalgard, MD PhD, Principal Investigator — Akerhus University Hospital
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

REFERENCES:
- [Derived] Lyngbakken MN, Berdal JE, Eskesen A, Kvale D, Olsen IC, Rueegg CS, Rangberg A, Jonassen CM, Omland T, Rosjo H, Dalgard O. A pragmatic randomized controlled trial reports lack of efficacy of hydroxychloroquine on coronavirus disease 2019 viral kinetics. Nat Commun. 2020 Oct 20;11(1):5284. doi: 10.1038/s41467-020-19056-6. PMID 33082342
- [Derived] Lyngbakken MN, Berdal JE, Eskesen A, Kvale D, Olsen IC, Rangberg A, Jonassen CM, Omland T, Rosjo H, Dalgard O. Norwegian Coronavirus Disease 2019 (NO COVID-19) Pragmatic Open label Study to assess early use of hydroxychloroquine sulphate in moderately severe hospitalised patients with coronavirus disease 2019: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jun 5;21(1):485. doi: 10.1186/s13063-020-04420-0. PMID 32503662